CLINICAL TRIAL: NCT00006101
Title: Randomized Placebo-Controlled, Double-Blind Phase IIb Chemoprevention Trial of Difluoromethylornithine in Brothers and First Cousin Males of Familial Prostate Cancer Probands
Brief Title: Eflornithine in Treating Patients At High Risk of Developing Prostate Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Thomas E. Ahlering (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor-Investigator, Thomas E. Ahlering, Professor, University of California, Irvine
Organization: University of California, Irvine (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: UCI 97-18 CDR0000068110; U01CA8188601 (Other: NCI); NCI-P00-0164 (Other: NCI); NCI-2009-00890 (Other: NCI Clinical Trials Reporting Program)
Record Dates: First submitted 2000-08-03; First posted 2003-01-27 (Estimated); Results first posted 2018-04-12 (Actual); Last update posted 2018-05-14 (Actual); Status verified 2018-04

CONDITIONS: Prostate Cancer
Keywords: stage I prostate cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Eflornithine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- eflornithine (Experimental): 500mg/d for 12 months
  Interventions: Drug: eflornithine
- Placebo (Placebo Comparator): placebo for 12 months
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: eflornithine — Take 500mg of DFMO per day for 12 months
  Other Names: Difluoromethylornithine (DFMO)
  Arms: eflornithine
Drug: Placebo — Take placebo per day for 12 months
  Arms: Placebo

SUMMARY:
RATIONALE: Chemoprevention therapy is the use of certain drugs to try to prevent the development of cancer. The use of eflornithine (DMFO) may be an effective way to prevent the development of prostate cancer.

PURPOSE: Randomized phase II trial to determine the effectiveness of eflornithine in preventing prostate cancer in patients who are at high risk of developing the disease.

DETAILED DESCRIPTION:
OBJECTIVES:

* Compare the levels of polyamines (putrescine, spermidine, and spermine) and progression-related genes in the prostate tissue of patients at high genetic risk for prostate cancer treated with eflornithine (DFMO) vs placebo.
* Determine the side effects of DFMO and compare them with the biological effect on the prostate gland in these patients.

OUTLINE: This is a randomized, double-blind, placebo-controlled study. Patients are stratified according to age (35 to 60 vs 61 to 70) and presence of localized cancer (yes vs no).

All patients receive oral placebo daily for 4 weeks. Patients who are compliant and take the placebo 5-7 days each week are randomized to one of two arms.

* Arm I: Patients receive oral placebo daily.
* Arm II: Patients receive high-dose oral eflornithine (DFMO) daily. Treatment continues for 1 year in the absence of unacceptable toxicity.

PROJECTED ACCRUAL: A total of 100 patients (50 per arm) will be accrued for this study within 3 years.

ELIGIBILITY:
Criteria for Eligibility

1. Men between the ages of 35 and 70 with family history of prostate cancer, i.e., prostate cancer diagnosed in two first degree relatives before the age of 70 years. (First degree relatives include a brother, father, and son.) There will be occasions in which a second or even third degree relative will be eligible. Additional information regarding these criteria is provided below and in Attachment 1.)

   * Two or more affected relatives of which at least 1 is a first degree relative or
   * At least two affected relatives, both of which are at least a second degree relative or
   * One first degree relative diagnosed with prostate cancer at age 55 or less.
2. No history of invasive cancer within 5 years (though non-melanoma skin or papillary bladder cancer will not be reason to exclude a patient); no prior history of prostate cancer, no severe metabolic disorders or other life-threatening acute or chronic disease; no additional x-ray or chemotherapy anticipated.

   * Men found to have localized prostate cancer (Gleason score ≤7) as part of the screening for the current trial, and opt for watchful waiting as their standard of care treatment for their condition, will be eligible to sign an additional consent form to continue with the randomization and on-study activities of this trial. On-study activities for these individuals will not differ from the on-study activities for the other men enrolled in this trial.
3. Must not require a medically mandated special diet which precludes compliance with study requirements
4. Not requiring regular use of anticoagulants on a regular basis. Prior use of chemoprevention agent(s) (such as Proscar) is allowed as long as the subject has been off the agent(s) for at least 3 months. Not currently participating in another prostate prevention trial.
5. Absence of history of current documented or symptomatic gastric or duodenal ulcer within 12 months prior to study entry, or of significant kidney or liver disease. No chronic anemia (hematocrit < 35 volume %), leukopenia (WEB <4,000) with normal differential, or thrombocytopenia (platelets <100,000) and with serum creatinine <1.5 mg/dl, serum bilirubin <2.0 mg/dl, and serum glutamic oxaloacetic transaminase (SGOT) or serum glutamic pyruvic transaminase (SGPT) <2× normal. Urinalysis should have <1+ protein, 0-3 casts, 0-5 white blood cell count (WBC) and red blood cell count (RBC).
6. Absence of any condition that predisposes to difficulties with hearing, wound healing or repair.
7. Must meet Southwest Oncology Group performance status criteria of 0-1 (0 = fully active, able to carry on all predisease activities without restriction [Karnofsky scale 90-100]; 1 = restricted in physically strenuous activity, but ambulatory and able to carry out work of a light or sedentary nature, i.e., light housework or office work [Karnofsky scale 70-80].
8. Subjects must be willing and able to keep required visits for study procedures and to complete study questionnaires.
9. Patient must not have had radiation therapy in the pelvic area.

Ages: 35 Years to 70 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Actual)
Dates: Start 1998-10; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Ahlering, MD, Principal Investigator — Professor
Locations (1):
- Chao Family Comprehensive Cancer Center at University of California Irvine Cancer Center, Orange, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Simoneau AR, Gerner EW, Nagle R, Ziogas A, Fujikawa-Brooks S, Yerushalmi H, Ahlering TE, Lieberman R, McLaren CE, Anton-Culver H, Meyskens FL Jr. The effect of difluoromethylornithine on decreasing prostate size and polyamines in men: results of a year-long phase IIb randomized placebo-controlled chemoprevention trial. Cancer Epidemiol Biomarkers Prev. 2008 Feb;17(2):292-9. doi: 10.1158/1055-9965.EPI-07-0658. PMID 18268112

RESULTS

PARTICIPANT FLOW:
Groups:
- Eflornithine: 500mg/d for 12 months
  eflornithine: Take 500mg of eflornithine (Difluoromethylornithine) per day for 12 months
Period: Overall Study
Arm/Group | Eflornithine | Placebo
Started | 38 | 38
Completed | 33 | 33
Not Completed | 5 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Eflornithine | Placebo | Total
Number analyzed (Participants) | 38 | 38 | 76
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 34 | 33 | 67
  >=65 years | 4 | 5 | 9
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 38 | 38 | 76
Region of Enrollment [Number; unit: participants]
  United States | 38 | 38 | 76

OUTCOME MEASURES:

1. Primary Outcome: Change in Total PSA, Percent Free PSA, and Prostate Volume at 12 Months
Description: Difference refers to absolute difference of 12 months to baseline and % relative difference refers to the ratio of the absolute difference divided by the baseline times 100.
Time Frame: Baseline and 12 months
Population: The results reported include all men with both an entrance and exit biopsy, regardless of cancer status.
Measure: Mean (Standard Deviation); unit: Relative % difference
Arm/Group | Eflornithine | Placebo
Number analyzed (Participants) | 34 | 33
Relative % difference
  Total PSA | -0.75 (26.29) | 1.55 (38.29)
  Percent Free PSA | 10.21 (44.39) | 4.89 (40.14)
  Prostate Volume | 0.94 (17.58) | 11.14 (19.44)

ADVERSE EVENTS:
Time Frame: Through study completion, an average of 1 year
Arm/Group | Eflornithine | Placebo
All-Cause Mortality (participants affected / at risk) | 0/38 | 0/38
Serious Adverse Events (participants affected / at risk) | 4/38 | 1/38
Other Adverse Events (participants affected / at risk) | 20/38 | 18/38
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Eflornithine (N=38) | Placebo (N=38)
Prostate Cancer Diagnosis (Reproductive system and breast disorders) | 3 | 1 — Diagnosed at 6 or 12 month biopsy
Knee Replacement (Surgical and medical procedures) | 1 | 0 — Hospitalized for full knee replacement
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Eflornithine (N=38) | Placebo (N=38)
Muscular skeletal complaints (Musculoskeletal and connective tissue disorders) | 7 | 2 — Complaints include disk disease, tendonitis, etc.
Hearing Related Complaints (Nervous system disorders) | 5 | 6 — Include tinnitus, vertigo, and hearing changes
Rash (Skin and subcutaneous tissue disorders) | 0 | 1
Chest Pain (General disorders) | 0 | 1
Vomiting (General disorders) | 0 | 1
Sexual Difficulties (Reproductive system and breast disorders) | 3 | 2
Gastrointestinal Side Effects (Gastrointestinal disorders) | 4 | 4
Flu or cold symptoms (General disorders) | 1 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No